CLINICAL TRIAL: NCT07227883
Title: Blinded, Randomized, Controlled, Trial to Evaluate the Efficacy and Safety of Autologous Hair Follicle Secretome for Facial Rejuvenation
Brief Title: Secretome Treatment for Facial Rejuvenation
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Acorn Biolabs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACN-301
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Facial Aging; Rejuvenation; Stem Cell; Stem Cell Banking
Keywords: stem cells; secretome; autologous; hair follicle; aging; facial; face; under eyes; wrinkles; anti-aging; rejuvenation; regeneration
MeSH Terms: conditions — Facies

STUDY DESIGN:
Intervention Model Description: Optional cross-over after blinded phase of study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor, except for clinical study managers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Saline will act as a control and will be intradermally injected.
  Interventions: Other: Control Saline
- Active-Secretome (Experimental): Autologous Hair follicle Derived Secretome
  Interventions: Other: Autologous Hair Follicle-Derived Secretome

INTERVENTIONS:
Other: Autologous Hair Follicle-Derived Secretome — This interventional product is a secretome derived from the stem cells that reside in the hair follicle.
  Other Names: aHFS; Hair Follicle Secretome; Hair Follicle Stem Cell
  Arms: Active-Secretome
Other: Control Saline — Saline solution will be the placebo control. The active is diluted with saline so this is an appropriate control.
  Arms: Control

SUMMARY:
Secretome treatment for facial rejuvenation

DETAILED DESCRIPTION:
This study will quantitatively evaluate the efficacy and safety of the autologous hair follicle secretome for skin rejuvenation. The secretome is produced by non-invasively collecting hair follicles by plucking 50-75 hairs. Ten follicles are selected to cultured in media (proprietary xeno- and human protein free) for 4 weeks and conditioned media is collected and lyophilized to produce the autologous secretome product. The secretome contains growth factors, extracellular matrix molecules, cytokines, exosomes, etc. Upon use, the autologous secretome is diluted in saline and used on the subject the hairs were collected from. This study is evaluating the efficacy and safety of intradermal injections of the secretome for facial rejuvenation. The study is a double-blind and open label extension phases, randomized, placebo-controlled trial. Double-blind up to 120 days, followed by an open label extension for control patients opting to cross-over and receive active treatment.

ELIGIBILITY:
Inclusion Criteria

* Male or Female
* Age: ≥30 and ≤ 75 at the time of consent.
* Fitzpatrick skin types I-V
* Moderate to very severe facial aging according to the SASSQ for the categories of elasticity, wrinkles, and skin roughness.
* Willing to refrain from cosmetic procedures throughout the study period (i.e. laser treatments, chemical peels, microneedling, dermal filler injections, neuromodulator injections, etc.)
* Willing to use study support products as directed and will not introduce any new skin care or makeup products throughout the study period. Subjects will be provided with a Skincare Kit: Cetaphil Gentle Skin Cleanser 20 oz, Cetaphil Daily Hydrating Lotion 3 oz, Cetaphil Sheer Mineral Liquid Face Sunscreen SPF 50 . Two of each will be provided with application instructions.
* Male subjects with facial hair must be willing to shave the morning of their treatments/follow-up visits.
* Willing to minimize sun/ultraviolet light exposure for the duration of the study, including all of the following: applying sunscreen daily, at least 15 minutes before going outside; wearing sun-protective clothing (e.g., a hat, sunglasses) when outdoors; reapplying sunscreen every 2 hours during outdoor activities; avoiding tanning bed/tanning product use.
* Competent and willing to provide written, informed consent to participate in all study activities
* Willing and able to tolerate multiple injections and attend all study visits
* Negative urine pregnancy test result at the time of screening (if applicable)
* For female subjects of childbearing potential, must be willing to use an acceptable form of birth control (oral contraceptives, hormonal implants, intrauterine device [IUD], hormonal injectables specifically for birth control, contraceptive patch or ring, tubal ligation [tubes tied], or total sexual abstinence) during the entire course of the study. All systemic birth control measures (oral, hormonal implants, injectables) must be in consistent use for at least 30 days prior to study enrollment. A female is considered of childbearing potential unless she is postmenopausal, without a uterus and/or both ovaries, or has had a bilateral tubal ligation.

Exclusion Criteria

* Use of topical tretinoin, adapalene, tazarotene, hydroquinone, imiquimod, 5-fluorouracil, ingenol mebutate, concentrated hydrogen peroxide, diclofenac, vitamin C, alpha hydroxy acids, or photodynamic therapy (PDT) to the face within 4 weeks prior to baseline photography and throughout the study period
* Dermatologic diseases or conditions (e.g. atopic dermatitis, psoriasis, rosacea, seborrheic dermatitis, wounds, infections, irritation, sunburn, windburn, etc.) in the treatment area that could interfere with the study, in the opinion of the Investigator
* Starting use or stopping use of GLP-1 agonists, or planned weight loss or gain during the study period. Subjects using GLP-1 agonists must be taking the drug for maintenance AND body weight must have been stable for at least 3 months prior to initial study treatment.
* History of keloid formation, hypertrophic scarring, or abnormal/delayed wound healing
* Previous medical aesthetic rejuvenation treatments on the face, such as chemical peel, dermabrasion, non-ablative or ablative resurfacing procedure, or face-lift with laser or other devices, up to 3 months prior to baseline photography
* Treatment with neuromodulators in crow's feet, glabellar region, or frontalis muscles within 4 months prior to baseline photography
* Treatment with dermal fillers, collagen stimulators, fat injections or permanent fillers within the past 6 months prior to baseline photography.
* Patients using other anti-aging treatments/procedures/systemic medications or injections administered/prescribed by a medical professional before starting the study, if the investigator believes they will confound the results. Consulting with Sponsor is encouraged.
* Heavy smoker (>1 pack of cigarettes a day)
* Energy-based device (i.e., radiofrequency device treatments, microfocused ultrasound device or other ultrasound-based device treatments, laser and light-based device treatments, microneedling) treatment in the treatment area within 6 months prior to baseline photography
* Currently be taking isotretinoin (Accutane).
* Subjects on an immunosuppressant or have an autoimmune condition (except stable, controlled Hashimoto's thyroiditis)
* Surgery (i.e., face lift, eyebrow lift, neck lift or lower rhytidectomy, liposuction, etc.) during the 12-month period prior to baseline photography
* Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
* Severe active infection (e.g. HIV, HepB or C, UTI, etc.)
* Current or recent (within last 5 years) malignancy (except basal cell and squamous cell skin cancers as long as basal cell was not on the face)
* History of systemic chemotherapy or radiation within the last 5 years
* Continuous/daily use of nonsteroidal anti-inflammatory or Vitamin E, unless discontinued within 7 days before 1st treatment and only used as needed through the trial period.
* Anticipated pregnancy or trying to become pregnant in the next year
* Current anticoagulant therapy (heparins; factor Xa inhibitors; direct agents such dabigatran, rivaroxaban, apixaban, endoxaban and betrixaban; warfarin/coumarins). Low dose aspirin and omega-3 supplements allowed.
* Any other criterion that is based on the clinical judgment of the investigator may place the subject at risk or confound study results

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline to 120days
  Adverse events and expected treatment effects will be collected at each time point. Spontaneously reported adverse events will also be collected.
VISIA-CR Skin Quality Scores (VISIA-CR is not an acronym, it is a brand name of the system) | Baseline, 30, 60, 90 and 120 days
  VISIA-CR photography and analysis of skin quality (redness, wrinkles, UV spots, skin roughness). Scores range from 0-100. Lower scores are improvement.

SECONDARY OUTCOMES:
Subject Satisfaction | 30, 60, 90 and 120 days
  Subject Satisfaction Scale is a 5-point Likert Scale. The scale is Dissatisfied, Neither Satisfied or Dissatisfied, Slightly Satisfied, Satisfied and Very Satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Steve Yoelin, MD, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No